CLINICAL TRIAL: NCT01097785
Title: Targeting Sympathetic Overactivity in Heart Failure Patients With Statins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-1135098
Record Dates: First submitted 2010-03-26; First posted 2010-04-02 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Active Comparator): 40 mg Simvastatin 1 pill every day for 30 days
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo cap 1 pill every day for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — 40 mg, P.O.,daily for 30 days
  Other Names: Zocor
  Arms: Simvastatin
Drug: Placebo — 1 capsule daily for 30 days
  Arms: Placebo

SUMMARY:
Heart failure (HF) is a leading cause of morbidity and mortality in the United States with the incidence and prevalence of the disease on a continual rise. An overactive sympathetic nervous system has become a hallmark characteristic of HF. Although sympathetic activation is initially beneficial to maintain cardiac output, blood pressure and perfusion to vital organs, over the long term it becomes deleterious contributing to the worsening of HF and sudden cardiac death. Indeed, recent findings in HF patients suggest that the sympathetic overactivity is not just a marker of poor prognosis but it plays a causative role in the development of the disease. Thus, the sympathetic nervous system constitutes a putative drug target in the treatment of HF. However, despite aggressive medical management, including conventional anti-adrenergic strategies, sympathetic nerve activity (SNA) has been shown to remain abnormally high in HF patients and improvements in survival have been limited. Thus, other treatment strategies that include reducing SNA and its deleterious consequences are warranted. Recent findings from clinical trials indicate that 3-hydroxy-3-methyl-glutaryl coenzyme A reductase inhibitors (statins) improve survival irrespective of cholesterol lowering bringing the pleiotropic (i.e., cholesterol independent) effects of statins to the forefront. An important pleiotropic effect recently reported in experimental HF, that has yet to be directly tested in human HF, is the ability of statins to reduce resting sympathetic outflow. Several studies in pacing-induced HF rabbits have demonstrated that statins normalize the excessive sympathetic activation in the HF state. Thus, the goal of this project is to determine whether these findings in experimental HF can be translated to the clinical setting of human HF. Our central hypothesis is that statins reduce sympathetic overactivity in HF patients. To test this hypothesis we will directly measure muscle SNA and perform a randomized crossover placebo control study. Subjects will come to the research laboratory before and after the administration of Simvastatin at a standard therapeutic dosage of 40 mg. per day or placebo for 1 month

DETAILED DESCRIPTION:
Heart failure (HF) is a leading cause of morbidity and mortality in the United States with the incidence and prevalence of the disease on a continual rise. An overactive sympathetic nervous system has become a hallmark characteristic of HF. Although sympathetic activation is initially beneficial to maintain cardiac output, blood pressure and perfusion to vital organs, over the long term it becomes deleterious contributing to the worsening of HF and sudden cardiac death. Indeed, recent findings in HF patients suggest that the sympathetic overactivity is not just a marker of poor prognosis but it plays a causative role in the development of the disease. Thus, the sympathetic nervous system constitutes a putative drug target in the treatment of HF. However, despite aggressive medical management, including conventional anti-adrenergic strategies, sympathetic nerve activity (SNA) has been shown to remain abnormally high in HF patients and improvements in survival have been limited. Thus, other treatment strategies that include reducing SNA and its deleterious consequences are warranted. Recent findings from clinical trials indicate that 3-hydroxy-3-methyl-glutaryl coenzyme A reductase inhibitors (statins) improve survival irrespective of cholesterol lowering bringing the pleiotropic (i.e., cholesterol independent) effects of statins to the forefront. An important pleiotropic effect recently reported in experimental HF, that has yet to be directly tested in human HF, is the ability of statins to reduce resting sympathetic outflow. Several studies in pacing-induced HF rabbits have demonstrated that statins normalize the excessive sympathetic activation in the HF state. Thus, the goal of this proposal is to determine whether these findings in experimental HF can be translated to the clinical setting of human HF. Our central hypothesis is that statins reduce sympathetic overactivity in HF patients. To test this hypothesis we will directly measure muscle SNA before and after one month of statin therapy. In addition, to begin to elucidate the potential mechanism(s) involved in statin-induced reductions in SNA we will use the technique of partial autospectral analysis to assess the baroreflex-independent (i.e., central) component of SNA and the application of neck pressure and neck suction to assess the baroreflex-dependent control of SNA. The significance of the proposed experiments is the potential of statin therapy to reduce SNA in HF patients providing a novel therapeutic strategy to target the heightened resting sympathetic drive present in HF.

The study will utilize a randomized crossover placebo-controlled study design. Subjects will come to the research laboratory before, during and after the administration of either a placebo or Simvastatin for one month at a standard therapeutic dosage of 40 mg per day. Subjects will be carefully monitored for any adverse effects by examining blood samples at baseline and 4 weeks for markers of liver, kidney, or muscle damage. If the subject's responses to one month of Simvastatin therapy are minimal, such that the decrease in LDL cholesterol is less than 25%, we will ask them to participate in an additional 2 weeks of Simvastatin administration at a dosage of 80 mg per day. During the baseline, the visit at 4 wks, and during the additional visit (if necessary) subjects will undergo the following experimental measurements and procedures, which will take approximately four hours. All measurements and procedures will be performed by the principal investigator and trained research personnel.

To completely obtain all the data necessary for this project, it would be expected to take 5 years. This is based on the goal of initially collecting additional data to add to the preliminary data of a recent American Heart Association (AHA) grant submission and then submitting the project for an NIH grant. Based on power calculations and previous experience using these experimental measures, it will take approximately 30 heart failure patients to determine the influence of statins on sympathetic nerve activity. This will permit statistical comparisons and takes into account the technical difficulties of obtaining repeat quality sympathetic nerve recordings in the same patient as well as the data collection necessary to determine the potential contribution of baroreflex-dependent and -independent mechanisms. Healthy control subjects matched to each HF patients for age, sex, and body mass index, all of which are known factors that influence resting SNA, will also be studied. These studies are important for comparison to determine whether these statin-induced reductions in SNA specific to HF or a general overall effect of statin therapy. It is anticipated that identifying patients not already on statin therapy may take some time as this therapy is standard in this patients group. We chose Simvastatin for our studies because this was the statin of choice in the pacing-induced HF rabbit studies that have reported a normalization of resting SNA after statin therapy. We anticipate that future studies identifying the efficacy of different statins in reducing SNA, the impact of different dosages, and different durations of treatment will be warranted.

ELIGIBILITY:
Inclusion Criteria:

* Male and females of all ethnic backgrounds ranging aged 18 to 70
* Ages 18-70 yrs
* Patients with congestive heart failure diagnosed on clinical history, a routine exercise test, echocardiography and/or routine cardiac catheterization, in functional class I-III
* Patients with heart failure due to ischemic and non-ischemic etiologies
* Normotensive and not taking blood pressure controlling medications

Exclusion Criteria:

* Low blood pressure (<100/60)
* End stage renal disease
* Chronic Obstructive Pulmonary Disease (COPD) with concurrent daily use of inhalers
* Peripheral neuropathy
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Fadel, PhD, Principal Investigator — University of Missouri-Columbia; Anand Chockalingam, M.D., Study Chair — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants were recruited; 6 were allocated to each arm.
Groups:
- Simvastatin, Then Placebo: Cycle 1: Participants received 40 mg Simvastatin 1 pill every day for 30 days. Cycle 2: Two week washout period. Cycle 3: Placebo pill once every day for 30 days.
- Placebo, Then Simvastatin: Cycle 1: Participants received Placebo capsule 1 pill every day for 30 days. Cycle 2: Two week washout period. Cycle 3: Simvastatin 40mg once every day for 30 days.
Period: Cycle 1 (30 Days)
Arm/Group | Simvastatin, Then Placebo | Placebo, Then Simvastatin
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Simvastatin, Then Placebo | Placebo, Then Simvastatin
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Cycle 3 (30 Days)
Arm/Group | Simvastatin, Then Placebo | Placebo, Then Simvastatin
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Quality muscle sympathteic nerve activity recordings obtained in 6 patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin, Then Placebo | Placebo, Then Simvastatin | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (3) | 51 (3) | 51 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 5 | 10
Muscle Sympathetic Nerve Activity [Mean (Standard Deviation); unit: bursts/100 heartbeats] | 45 (14) | 59 (13) | 52 (14)

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Sympathetic Nerve Activity in Bursts Per 100 Heartbeats
Description: Muscle sympathetic nerve activity will be assessed after one month of placebo and statin therapy; measured in bursts/100 heartbeats.
Time Frame: Baseline and 30 days
Measure: Mean (Standard Error); unit: bursts/100 heartbeats
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 12 | 12
bursts/100 heartbeats | 59 (5) | 45 (6)
Statistical Analysis 1: Comparison: Simvastatin vs Placebo; Test type: Superiority or Other; p < 0.05, Student's t-test

2. Secondary Outcome: Change in Measures of Reactive Oxygen Species in the Blood
Description: Reactive Oxygen Species will be assessed after one month of placebo and statin therapy; measured using electron parametric resonance spectroscopy (EPR).
Time Frame: Baseline and 30 days
Measure: Mean (Standard Error); unit: EPR Arbitrary Units
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 12 | 12
EPR Arbitrary Units | 8671500.00 (1584626.44) | 14056500.00 (1010765.39)
Statistical Analysis 1: Comparison: Simvastatin vs Placebo; Test type: Superiority or Other; p < 0.05, Student's t-test

ADVERSE EVENTS:
Arm/Group | Simvastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No